CLINICAL TRIAL: NCT06267300
Title: Treatment of Post-COVID-19 With Hyperbaric Oxygen Therapy: a Randomized, Controlled Trial
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Da Vinci Clinic (Unknown); HGC Rijswijk (Unknown)
Responsible Party: Principal Investigator, Merel Hellemons, Dr., Erasmus Medical Center
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Record Dates: First submitted 2024-02-19; First posted 2024-02-20 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Post-COVID-19 Syndrome; Post-COVID Syndrome; Post COVID-19 Condition; Post-COVID Condition; Post COVID-19 Condition, Unspecified; Long COVID; Long Covid19
Keywords: clinical relevance; quality of life; absence from work; cost-effectiveness
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial comparing HBOT to standard care alone, with a cross-over from standard care to HBOT in case primary outcome is positive after 6 months follow-up.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hyperbaric Oxygen therapy (Experimental): 40 sessions of HBOT at 2.4 ATM
  Interventions: Drug: Hyperbaric oxygen
- Standard care (No Intervention)

INTERVENTIONS:
Drug: Hyperbaric oxygen — Hyperbaric oxygen therapy (2.4 ATA, 40 sessions)
  Other Names: HBO; HBOT; Hyperbaric oxygen therapy
  Arms: Hyperbaric Oxygen therapy

SUMMARY:
The goal of this clinical try is to investigate the effect of hyperbaric oxygen therapy (HBOT) on symptoms, quality of life and absence of work through sickness in patients with post-COVID on short- and mid-term, as well as to identify biochemical mechanisms of action.

The main questions it aims to answer are:

* What is the clinical relevance of improvements of symptoms and quality of life after treatment with HBOT for post-COVID?
* What are the changes in absence from work after treatment with HBOT?
* What is the cost-effectiveness of treatment with HBOT?
* What are possible mechanisms of action of HBOT?

Participants will undergo 40 sessions of HBOT. Researchers will compare HBOT with standard care alone (control group). In case of a positive outcome, patients in the control group can cross-over to the HBOT group after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Cognitive and/or physical symptoms ≥ 12 months after acute COVID-19 infection
* Symptoms include post-exertional malaise (PEM) and/or dysautonomia as assessed by questionnaires and/or NASA LEAN test
* Symptoms affect day-to-day life (based on SF-36 'role limitations due to physical functioning' score of ≤ 50 at baseline).
* Current treatment regimen is stable for at least 1 months before inclusion

Exclusion Criteria:

* Unfit for hyperbaric treatment
* Previous diagnosis of ME/CFS
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Physical and mental component scores of the 36-item Short Form Survey (SF-36) | Week 20 (i.e. 3-months after end of HBOT)
  Range 0-100, with higher scores indicating higher quality of life

SECONDARY OUTCOMES:
Euroqol-5D (EQ-5D) | Week 0/4/8/20/34 (i.e. at start of HBOT, halfway during treatment, directly after treatment and 3 and 6 months after treatment).
  Descriptive for 5 dimensions + visual analogue score (VAS, range 0-100 with higher scores indicating higher quality of life)
Activity tracking (through wrist band), monitoring heart rate, step count and sleep patterns | Worn continuously until week 34
Biochemical parameters | Week 0, 8 and 34 (i.e. at start of HBOT, directly after HBO and 3-months after treatment)
Absence from work | Week 0/4/8/20/34 (i.e. at start of HBOT, halfway during treatment, directly after treatment and 3 and 6 months after treatment).
Cost-effectiveness | Week 0/4/20/34 (i.e. at start of HBOT, directly after treatment and 3 and 6 months after treatment).

CONTACTS AND LOCATIONS:
Locations (7):
- Netherlands (7):
  - Da Vinci Clinic, Amersfoort
  - Da Vinci Clinic, Geldrop
  - Da Vinci Clinic, Hoogeveen
  - HGC Rijswijk, Rijswijk
  - Da Vinci Clinic, Rotterdam
  - Erasmus MC, Rotterdam
  - Da Vinci Clinic, Waalwijk